CLINICAL TRIAL: NCT04079673
Title: The Effect of Perioperative Epidural Anesthesia and Analgesia on Gut Microbiota and Gastrointestinal Function Recovery in Living Donor Hepatectomy
Brief Title: Perioperative Epidural Anesthesia and Analgesia on Gut Microbiota
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 201812090RINC
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2020-10

CONDITIONS: Living Donor Hepatectomy
Keywords: epidural anesthesia; microbiota
MeSH Terms: interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient controlled epidural analgesia (Active Comparator): Use of patient controlled epidural analgesia (PCEA) for postoperative pain control
  Interventions: Procedure: Patient controlled epidural analgesia
- Intravenous patient controlled analgesia (Sham Comparator): Use of intravenous patient controlled analgesia(IVPCA) for postoperative pain control
  Interventions: Drug: Intravenous patient controlled analgesia

INTERVENTIONS:
Procedure: Patient controlled epidural analgesia — Patient controlled epidural analgesia with marcaine 0.66mg/ml +fentanyl 1.75mcg/ml for postoperative pain control
  Other Names: PCEA
  Arms: Patient controlled epidural analgesia
Drug: Intravenous patient controlled analgesia — Intravenous patient controlled analgesia with morphine 1mg/ml for postoperative pain control
  Other Names: IVPCA
  Arms: Intravenous patient controlled analgesia

SUMMARY:
As the only curative treatment for end-stage liver diseases, liver transplantation has been widely carried out around the world. The shortage of organs from deceased donors facilitate the adoption of living donor liver transplantation. Living donor hepatectomy is the most massive operation a healthy person could undergo, so donor safety is of utmost importance. However, previous studies focused on the outcomes of liver transplant recipients. There are still many uncertainties about the recovery in living liver donors.

The body microorganisms that reside in the human intestinal tract, referred to as the gut microbiota, are essential to human metabolism and immunity. The physiological functions of microbiota include defense against pathogens, providing nutrients such as vitamin B12 folate and vitamin K, and modulating gut integrity and permeability. Despite relatively stable microbiota during life, different illnesses, surgeries, medications dietary factors, and lifestyle changes could contribute to the imbalance of ecosystems resulting many gastrointestinal and extra-gastrointestinal disorders. Many researches have established a relationship between the gut microbiome and patients with liver disease such as liver cirrhosis, alcoholic liver disease and obesity related liver diseases etc. These liver disorders are associated with bacterial overgrowth, dysbiosis, and increased intestinal permeability. However, the relationship between hepatectomy and microbiota has not been fully investigated, especially in healthy liver donors.

Many routine perioperative management can impact the state of the microbiome and therefore can impact clinical outcomes, like bowel preparation and antibiotics. Potential factors affecting the gut microbiota also include perioperative manipulation, stress released hormones, and opioids. Maintenance of proper anesthetic depth is beneficial to attenuate surgical stress. However, general anesthesia including volatile anesthetics and opioids, is associated with altered gut microbiota. Therefore, regional anesthesia and analgesia which effectively attenuating surgical stress while efficiently reducing general anesthetics consumption, seem to provide promising advantages. Epidural analgesia has been proved to improve gastrointestinal function in major abdominal and thoracic surgery. However, the effect of perioperative epidural anesthesia and analgesia on microbiota is not clear.

ELIGIBILITY:
Inclusion Criteria:

1. Expected to receive living liver hepatectomy in National Taiwan University Hospital, age between 20 and 55 years old.

Exclusion Criteria:

1. Previous use of antibiotics within four weeks.
2. Previous gastrointestinal surgery.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-19 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Microbiota analysis | one month
  16S metagenomic sequence processing

SECONDARY OUTCOMES:
LPS-binding protein | one month
  LPS-binding protein(mcg/mL)
Intestinal fatty acid binding protein | one month
  Intestinal fatty acid binding protein(ng/mL)
IgA | one month
  IgA(mcg/mL)
IL-6 | one month
  IL-6(ng/mL)
I-FEED scoring | one week
  I-FEED scoring system for postoperative gastrointestinal function:
  1. Intake(score): tolerating oral diet(0), limited tolerance(1), complete Intolerance(3)
  2. Feeling nauseated(score): none(0), responsive to treatment(1), resistant to treatment(3)
  3. Emesis(score): none(0), ≧1 episode of low volume(<100mL) and none bilious(1), ≧1 episode of high volume(>100mL) or bilious(3)
  4. Exam(score): no distension(0), distension without tympany(1), significant distension with tympany(3)
  5. Duration of symptoms(score):0-24hours(0),24-72hours(1),>72hours(2)
  Total score: 0-2 normal, 3-5 postoperative GI intolerance, >6 postoperative GI dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Kuang-Cheng Chan, M.D.,PhD, Principal Investigator — Department of Anesthesiology, Natioanal Taiwan University Hospital
Locations (1):
- Department of Anesthesiology, National Taiwan University Hospital, Taipei, Taiwan